CLINICAL TRIAL: NCT05072730
Title: Super High-Pressure Balloon Versus Intravascular Lithotripsy for Severely Calcified Coronary Lesions: The ComparIson of Strategies to PrepAre SeveRely CALCified Coronary Lesions (ISAR-CALC) 2 Randomized Trial
Brief Title: ComparIson of Strategies to PrepAre SeveRely CALCified Coronary Lesions 2
Acronym: ISAR-CALC2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Abbott Medical Devices (Industry); SIS Medical AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE Nr. BA00421
Record Dates: First submitted 2021-06-18; First posted 2021-10-11 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Calcified Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Super high-pressure balloon (OPN NC) (Experimental): Patients will be treated with a Super High Pressure percutaneous transluminal coronary angioplasty (PTCA) Balloon (OPN NC).
  Interventions: Device: Super High Pressure Balloon (OPN NC)
- Intravascular lithotripsy (IVL) (Experimental): Patients will be treated with intravascular lithotripsy (IVL).
  Interventions: Device: Intravascular lithotripsy (IVL)

INTERVENTIONS:
Device: Super High Pressure Balloon (OPN NC) — Strategy of super high-pressure balloon angioplasty after unsuccessful lesion preparation with conventional NC balloon angioplasty.
  Optical coherence tomography (OCT) imaging will be performed after lesion preparation with OPN balloon. Optional additional pre-dilatation with OPN/standard NC balloon is permitted at the operator´s discretion. Following lesion preparation, stenting will be performed in the same setting using a latest-generation everolimus-eluting stent (XIENCE; Abbott Vascular, Chicago, IL, USA). Optional post-dilatation with OPN balloon or standard NC balloon is permitted at the operator´s discretion.
  Arms: Super high-pressure balloon (OPN NC)
Device: Intravascular lithotripsy (IVL) — Strategy of IVL after unsuccessful lesion preparation with conventional NC balloon angioplasty.
  Optical coherence tomography (OCT) imaging will be performed after lesion preparation with IVL balloon. Optional additional pre-dilatation with standard NC balloon is permitted at the operator´s discretion. Following lesion preparation, stenting will be performed in the same setting using a latest-generation everolimus-eluting stent (XIENCE; Abbott Vascular, Chicago, IL, USA). Optional post-dilatation with standard NC balloon is permitted at the operator´s discretion.
  Arms: Intravascular lithotripsy (IVL)

SUMMARY:
The ISAR-CALC 2 trial is an investigator-initiated, prospective, randomized, multicenter, assessors-blind, open-label other clinical investigation. The objective of this trial is to investigate final angiographic minimal lumen diameter (MLD) following a strategy of super high-pressure balloon (OPN NC) versus intravascular lithotripsy (IVL) for drug-eluting stent (DES) implantation in severely calcified coronary lesions.

DETAILED DESCRIPTION:
Detailed information is provided elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years and able to give consent
* Persistent angina despite medical therapy and/or evidence of inducible ischemia
* De-novo lesion in a native coronary artery
* Target reference vessel diameter or intended stent diameter ≥2.50 or ≤4.00 mm by visual estimation
* Severe calcification of the target lesion as determined by visual estimation at coronary angiography
* Unsuccessful lesion preparation with standard non-compliant balloon (< 30% reduction of baseline diameter stenosis at maximal pressure)
* Written informed consent.

Exclusion Criteria:

* Target lesion is located in a coronary artery bypass graft
* Target lesion is an in-stent restenosis
* Target lesion is a chronic total occlusion
* Target vessel thrombus
* Limited long-term prognosis due to other comorbid conditions with life expectancy <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Final angiographic minimal lumen diameter | Intraprocedural.
  The primary outcome measure of the trial is the final angiographic minimal lumen diameter as assessed by angiographic core laboratory.

SECONDARY OUTCOMES:
Angiographic Success | Intraprocedural.
  Defined as target lesion residual angiographic stenosis < 30% in the presence of Thrombolysis in Myocardial Infarction (TIMI) 3 flow.
Procedural Success | During index hospitalization, assessed up to 30 days.
  Defined as angiographic success without the occurrence of major adverse cardiac event (MACE), a composite of cardiac death, target-vessel related MI and repeat target-vessel revascularization, during index hospitalization.
Strategy Success | Intraprocedural.
  Defined as procedural success using the assigned study device and DES, without requirement for additional devices for lesion preparation; i.e. rotational atherectomy
Acute lumen gain | Intraprocedural.
  Defined as minimal lumen diameter (MLD) after balloon angioplasty with the assigned study devices minus baseline MLD.
Complementary lesion preparation | Intraprocedural.
  Need for complementary lesion preparation with rotational atherectomy
MACE rates | 30 days.
  Occurrence of major adverse cardiac event (MACE) up to 30 days.
Stent expansion as assessed by OCT imaging. | Intraprocedural.
  Stent expansion index, defined as minimum stent area divided by mean reference lumen area assessed with OCT imaging.
Cost-effectiveness analysis | Intraprocedural.
  Cost-effectiveness analysis of OPN versus IVL in severely calcified coronary lesions treated with DES implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Cassese, MD, PhD, Principal Investigator — Deutsches Herzzentrum Munich; Tobias Rheude, MD, Principal Investigator — Deutsches Herzzentrum Munich
Locations (4):
- Germany (4):
  - Herz- und Diabeteszentrum NRW Universitätsklinikum der Ruhr-Universität Bochum, Bad Oeynhausen
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - MEDICLIN Herzzentrum Lahr, Lahr
  - Deutsches Herzzentrum Muenchen, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scalamogna M, Abdel-Wahab M, Mashayekhi K, Fusaro M, Leistner DM, Ayoub M, Xhepa E, Joner M, Kastrati A, Cassese S, Rheude T. Randomized ComparIson of Strategies to PrepAre SeveRely CALCified Coronary Lesions 2: Design and Rationale of the ISAR-CALC 2 Trial. Cardiovasc Revasc Med. 2023 Apr;49:22-27. doi: 10.1016/j.carrev.2022.12.008. Epub 2022 Dec 30. PMID 36609101